CLINICAL TRIAL: NCT03797625
Title: Endostar Combined With IP Second-line Treatment of Advanced Esophageal Squamous Cell Carcinomas of the Prospective, Single Arm Phase II Clinical Study
Brief Title: Endostar Combined With IP Second-line Treatment of Advanced Esophageal Squamous Cell Carcinomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-SH-002
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Irinotecan; Cisplatin; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endostar Combined With IP (Experimental): Endostar15mg/m2 Irinotecan 60mg/m2，D1，8 DDP 60mg/m2，D1
  Interventions: Drug: Irinotecan; Drug: DDP; Drug: Endostar

INTERVENTIONS:
Drug: Irinotecan — 60mg/m2，D1，8
Drug: DDP — 60mg/m2，D1
  Other Names: Cisplatin
Drug: Endostar — 15mg/d，d1-d7 civ
  Other Names: ENDO

SUMMARY:
The aim of this study is to explore whether endostar combined with IP as treatment could improve progression-free surial time (PFS) and to evaluate the safety of the chemotherapy regimens

DETAILED DESCRIPTION:
This study is to explore whether endostar combined with IP as treatment could improve progression-free surial time (PFS) and to evaluate the safety of the chemotherapy regimens used as second-line treatment of advanced esophageal squamous cell carcinomas

ELIGIBILITY:
Inclusion Criteria:

Histologically proven primary thoracic esophageal squamous cell carcinoma According to the esophageal AJCC2009 7th to determine new stage IV esophageal cancer The subject has PD after first-line chemotherapy or radiation within a year Presence of at least one index lesion measurable by CT scan or MRI according to RECIST 1.1 Can eat more than liquid diet; No signs before esophageal perforation 18~75 years PS:0-1 Life expectancy of ≥ 3 months ANC ≥ 2×109/L，PLT ≥ 100×109/L，Hb ≥ 90g/L TB ≤ UNL； ALT/AST ≤ 2.5×UNL，AKP ≤ 5×UNL Ccr≤ UNL,Scr≥60 mL/min Normal electrocardiogram (ecg), the body had no unheal wounds Radiotherapy before within the scope of the normal dose and not affect subsequent treatment Prior to biological agents, especially e. coli genetically engineered products without severe allergic reactions Signed written informed consent

Exclusion Criteria:

Breast-feeding or pregnant women, no effective contraception if risk of conception exists Chronic diarrhea, enteritis, intestine obstruction which are not under control Esophageal obstruction cannot eat liquid completely, esophagus have deep ulcer perforation or hematemesis; Esophageal cancer common complications such as anastomotic leakage, serious lung complications, etc.

A second primary tumor (except skin basal cell carcinoma) The original serious heart disease, including: higher risk of congestive heart failure, unable to control arrhythmia, unstable angina, myocardial infarction, severe valvular heart disease, and resistant hypertension With uncontrol nerve, mental illness or mental disorders, compliance is poor, can't cooperate with accounts and response to treatment; Primary brain tumors or CNS metastases illness did not get a control, has obvious cranial hypertension or nerve mental symptoms With bleeding tendency Has inherited bleeding evidence of physical or blood coagulation disorder With clear chemotherapy drug allergy Other researchers believe that patients should not participate in this testing

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Overall Officials: chang jian hua, PD, Principal Investigator — PI; wang hui jie, doctor, Principal Investigator — SUBI
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Z, Sun S, Zhao X, Yu H, Wu X, Wang J, Chang J, Wang H. Rh-Endostatin Plus Irinotecan/Cisplatin as Second-Line Therapy for Advanced Esophageal Squamous Cell Carcinoma: An Open-Label, Phase II Study. Oncologist. 2022 Apr 5;27(4):253-e312. doi: 10.1093/oncolo/oyab078. PMID 35380726